CLINICAL TRIAL: NCT01731535
Title: Evaluation of the Risk for Radiographic and Clinical Nonunion in Patients With Previous Bisphosphonates Therapy.
Status: Withdrawn | Type: Observational
Why Stopped: It was a project initiated by a trainee but did not progress to subject accrual.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0437
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Non-union or Delayed Healing Fractures
Keywords: osteoporosis, low trauma fracture, non-union fracture, delayed healing fracture, bisphosphonate
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures; Fractures, Ununited

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prior bisphosphonate users: Patients with record of using bisphosphonate medication

SUMMARY:
Dose and duration of bisphosphonate therapy will increase the likelihood that patients experience delayed healing of non-union fractures.

DETAILED DESCRIPTION:
We intend to review the UWHealth patient database to identify individuals with delayed or nonunion fractures. Subsequently, we will collect associated medical information related to fractures such as age of osteoporosis diagnosis, BMI, previous bisphosphonate treatment, type and location of fracture, time to complete union, other treatment needed for nonunion etc. With this information, we will evaluate the risk of delayed and nonunion fractures in patients previously receiving bisphosphonate treatment compared to a normal population. We also will investigate other potential causes of delayed or nonunion fractures in this population.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 60 years old with delayed or nonunion low trauma fracture between 01/01/2000 - 12/31/2011.

Exclusion Criteria:

* None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women older than 60 years old with delayed or nonunion low trauma fracture beween 01/01/2000 - 12/31/2011.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The number of patients with delayed healing or non-union fractures with prior bisphosphonate use | 01/01/2000 - 12/31/2011
  This variable will be generated by reviewing diagnosis codes from patients seen at the University of Wisconsin Hospital and Clinics during the time period identified above.

SECONDARY OUTCOMES:
Evaluation of patient variables (demographic or medical history) related to non-union or delayed healing fractures. | 1/1/2000-12-31-2012
  Patients with non-union or delayed healing fractures obtaining care at the University of Wisconsin Hospital or Clinics will have a medical record review conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States